CLINICAL TRIAL: NCT04741048
Title: A Pre-market, Open-label Feasibility, Prospective, Single-arm Multicenter Feasibility Investigation of Hearing Performance Using the CI624 in Adults With Low-frequency Residual Hearing.
Brief Title: Hearing Implant Performance in Adults With Low-Frequency Residual Hearing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to cancel the study prior to any subjects being enrolled/consented due to the lack of CMS coverage and an internal staffing shortage.
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CAM5777
Record Dates: First submitted 2021-01-10; First posted 2021-02-05 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Sensorineural Hearing Loss; Low-Frequency Residual Hearing
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CI624 Slim 20 Electrode (Experimental)
  Interventions: Device: CI624 Slim 20 Electrode

INTERVENTIONS:
Device: CI624 Slim 20 Electrode — Cochlear Ltd CI624 cochlear implant with Slim 20 Electrode

SUMMARY:
The purpose of the feasibility study is to investigate hearing performance (audiometry and speech perception) using the CI624 in a group of adults (n=15) with low-frequency residual hearing who meet inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years-of-age or older at the time of surgery.
2. Low-frequency threshold at 500 Hz ≤ 50 dB HL and high-frequency pure-tone average (PTA), 2000-8000 Hz ≥ 65 dB HL in the ear to be implanted.
3. Pure-tone average (PTA) (0.5k, 1k, 2k Hz) > 30 dB HL in the contralateral ear.
4. CNC word recognition scores (mean of two lists) ≤ 60% in the ear to be implanted and ≤ 80% in the contralateral ear.
5. English spoken as a primary language.
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Individuals older than 70 years at the time of surgery.
2. Duration of severe to profound sensorineural hearing loss > 20 years per self-report.
3. Onset of sensorineural hearing loss, for the purpose of this study, prior to 5 years-of-age.
4. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
5. Conductive overlay of 15 dB or greater at two or more frequencies, in the range of 250 through 1000 Hz in the ear to be implanted.
6. Hearing loss of neural or central origin.
7. Diagnosis of Auditory Neuropathy.
8. Active middle-ear infection.
9. Medical or psychological conditions that contraindicate undergoing surgery as determined by the Investigator.
10. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the device and/or procedure, as determined by the Investigator.
11. Additional handicaps that would prevent or restrict participation in the audiological evaluations as determined by the Investigator.
12. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
13. Investigator site personnel directly affiliated with this study and/or their immediate family (spouse, parent, child, or sibling).
14. Cochlear employees or employees of a Contract Research Organization (CRO) or contractors engaged by Cochlear for the purposes of this investigation.
15. Currently participating, or has participated in the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Characterize hearing performance of the CI624. | 14 months
  Hearing performance of the CI624 will characterized using Constant Nucleus Constant (CNC) word recognition in quiet. Performance is scored as percent correct words.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacksonville Hearing and Balance, Jacksonville, Florida, United States